CLINICAL TRIAL: NCT02736370
Title: Early Weight Bearing for Bimalleolar and Trimalleolar Ankle Fractures Without Syndesmotic Disruption
Brief Title: Early Weight Bearing for Ankle Fractures
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-081
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Broken Ankle
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to assess the rate of return to work, rate of return to activities, functional outcome measures and pain scores in operatively repaired rotational Bimalleolar and Trimalleolar (AO/OTA Classification of 44A and 44B) ankle fractures not requiring fixation of the syndesmosis and allowed early weight bearing on or before the first post-operative visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages of 18 and up
* Closed, low-energy Bimalleolar and Trimalleolar rotational ankle fractures
* Orthopaedic Trauma Association (OTA) classification of 44A and 44B
* English speaking
* Able and willing to consent

Exclusion Criteria:

* Open fractures
* OTA classification of 43 and 44C
* Patients with diabetes mellitus
* No other lower extremity injuries that would affect functional outcomes
* Previous use of walking aides
* Patients with paralysis or hemiplegia
* Ankle fractures requiring syndesmotic repair
* Ankle fractures requiring fixation of the posterior malleolar
* Associated neurovascular injury
* Problems maintaining follow up (homeless or not willing to return for follow up)
* Pathological fractures
* Prisoners
* Patients not allowed to bear weight before the 6 week post-operative follow up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present with bimalleolar or trimalleolar ankle fractures
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-05; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Functional Outcome Scores | 12 months post operatively
  During follow up visits functional outcomes scores will be assess using the Foot and Ankle Score and the PROMIS (Patient Reported Outcomes Measurement Information System) Mobility Measure questionnaires. These forms will be analyzed together to determine the patients functional outcomes.

SECONDARY OUTCOMES:
Return to work | up to 12 months
  During follow up visits the patients return to work status will be assessed.
Fracture Healing | up to 12 months
  During follow up visits fractures healing will be assessed by physician review of x-rays.
Pain Scores | 12 months post operatively
  Pain Scores and PROMIS Pain Intensity and Interference questionnaires will be assessed during follow up. These forms will be analyzed together to determine the patients overall pain.
Post operative complications | up to 12 months
  Post operative complications will be assessed during follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Blake W Miller, DO, Principal Investigator — Corewell Health West

IPD SHARING:
Plan to Share IPD: No